CLINICAL TRIAL: NCT00657111
Title: CS-8958 - A Phase I, Double-Blind, Placebo Controlled, Ascending Single Inhaled Dose, Safety, Tolerability and Pharmacokinetic Study in Elderly Subjects
Brief Title: CS-8958 Single Inhaled Dose in Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-0064; CCRU 1833-174
Record Dates: First submitted 2008-04-10; First posted 2008-04-14 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Influenza
Keywords: influenza, elderly, United Kingdom; Vaxart
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- A1 (Experimental): Subjects 01-08; 5 mg CS-8958
  Interventions: Drug: CS-8958 formulated as dry powder
- A2 (Placebo Comparator): Subjects 01-08; placebo
  Interventions: Other: Placebo
- B1 (Experimental): Subjects 09-16; 10 mg CS-8958
  Interventions: Drug: CS-8958 formulated as dry powder
- B2 (Placebo Comparator): Subjects 09-16; placebo
  Interventions: Other: Placebo
- C1 (Experimental): Subjects 17-24; 20 mg CS-8958
  Interventions: Drug: CS-8958 formulated as dry powder
- C2 (Placebo Comparator): Subjects 17-24; placebo
  Interventions: Other: Placebo
- D1 (Experimental): Subjects 25-32; 40mg CS-8958
  Interventions: Drug: CS-8958 formulated as dry powder
- D2 (Placebo Comparator): Subjects 25-32; placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CS-8958 formulated as dry powder — CS-8958, formulated as a dry-powder and will be administered from capsules containing 5 mg CS-8958 and lactose to 25 mg (placebo) inserted into a FlowCaps inhaler device.
  Arms: A1; B1; C1; D1
Other: Placebo — placebo capsules containing 25 mg lactose
  Arms: A2; B2; C2; D2

SUMMARY:
The purpose of this study is to test the safety and tolerability of an investigational inhaled flu medication, CS-8958. Study participants will include 38 elderly males and females, age 65 and older. Participants will be divided into 1 of 4 possible treatment groups (Groups A, B, C and D) to receive the study drug or placebo (substance containing no medication). Group A will receive 5 mg CS-8958, Group B will receive 10 mg CS-8958, Group C will receive 20 mg CS-8958 and Group D will receive 40mg CS-8958. Safety information will be reviewed prior to administering a higher dose of treatment. Study procedures will include blood and urine samples, ECGs (measure of heart activity), and a 7 day clinic stay. Participants will be involved in study related procedures for up to 6 weeks.

DETAILED DESCRIPTION:
Influenza is an acute febrile illness caused by influenza A and B virus affecting all age groups. Influenza occurs annually and each year it is estimated that influenza epidemics cause 36,000 deaths and 114,000 hospitalizations in the US alone. Influenza infections are generally self-limiting; however significant morbidity and mortality can occur, predominantly in high risk groups such as the elderly and those suffering from chronic conditions. This study is a Phase I, double-blind, placebo-controlled, ascending single inhaled dose, safety, tolerability and pharmacokinetic study in elderly subjects with stable health status. The primary objective of this study is to evaluate the safety and tolerability of CS-8958 (5, 10 20 and 40 mg) in elderly subjects after a single dose administered via inhalation. Primary outcome measures of safety and tolerability will be addressed in terms of occurrences of treatment-emergent adverse events (AEs), changes in vital signs including blood pressure and pulse rate, functional oxygen saturation of arterial hemoglobin, oral body temperature, electrocardiogram, spirometry [Forced Vital Capacity (FVC)], Forced Expiratory Volume in 1 second (FEV1), Forced Expiry Volume percentage in 1 second (FEV1.0%), Forced Expiratory Flow Rate (FEF) 25%-75%), Peak Expiratory Flow Rate (PEFR, also called PEF), physical examinations, psychological assessments, and laboratory parameters. The secondary objectives of this study are to assess the systemic exposure of CS-8958 and its active metabolite R-125489 after single inhaled doses of CS-8958 in elderly subjects. The secondary outcome measures of pharmacokinetic parameters will be calculated for CS-8958 and R-125489 (active metabolite) concentrations in plasma and urine using a non-compartmental approach. These measurements will be used to assess the systemic exposure of CS-8958 and its active metabolite in elderly subjects after a single inhaled dose of CS-8958 (5, 10, 20 and 40 mg). This data will help to determine safety margins for dosing of elderly subjects in future studies. Thirty-eight healthy adults (male and female), aged 65 years and older, with stable health status, will be recruited for this UK based study. Subjects will be studied in 4 groups (Groups A to D) with each group consisting of at least 8 subjects. Within each group, subjects will be randomly allocated to Arm 1 or Arm 2. Arm 1 will receive the investigational drug with lactose to 25 mg (placebo) and Arm 2 will receive placebo only. Treatment will begin with a low dose of 5 mg (Group A) and subsequent higher doses of 10, 20 and 40 mg (Group B, C and D, respectively) It is planned that doses will be administered in an escalating manner. The Safety Monitoring Committee will review the safety, tolerability and pharmacokinetic data from each group prior to administration of the next dose. Following these reviews, the dose increment for subsequent groups may be increased, or the doses administered may be reduced, and may be lower than the starting dose. The maximum dose level to be studied will be 40 mg. The duration of the study for each subject will be a maximum of 6 weeks from initial screen to the follow-up visit. The screening period will be at most 4 weeks followed by 7 days in the clinic and a follow up visit 5-7 days after leaving the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male and female adults aged 65 years and older.
* Elderly adults in good health, as determined by vital signs (heart rate less than 100 bpm, blood pressure [systolic less than or equal to 160 mm Hg and diastolic less than or equal to 90 mm Hg], oral temperature less than or equal to 37.7 degrees C and SpO2 of at least 95%), stable medical condition and a full physical examination. A stable medical condition is defined as no change in medication, dose, or frequency of medication in the last 1 month; health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months; and no unplanned hospitalizations within the last 3 months (hospitalizations for minor elective procedures may be considered for inclusion on a case by case basis following discussion between the Investigator and the DMID Medical Monitor).
* Female subjects must be surgically sterile or post-menopausal (defined by a measurement of follicle stimulating hormone [FSH] greater than 18 mlU/mL and serum oestradiol less than 110 pmol/L (or 30 pg/mL), or by 24 consecutive months of amenorrhoea for which there is no other obvious pathological cause) and have a negative serum pregnancy test.
* No clinically significant abnormality in the ECG. QTc must be less than 450 ms and PR 120-209 ms. Any ECGs considered abnormal will be reviewed and approved by an independent cardiologist, (normal variants such as sinus arrhythmia and sinus bradycardia do no need to be independently reviewed).
* Negative results in Human Immunodeficiency Virus (HIV) antibody, Hepatitis B surface antigen (HBsAg) and Hepatitis C antibody tests.
* Negative results in urine drug screen and alcohol breath test.
* Able to understand and comply with all planned study procedures including ability to perform respiratory testing and use the inhaler device after training.
* Provide informed consent prior to any study procedures and is available for all study visits.

Exclusion Criteria:

* A Grade 2 biochemistry, hematology or urinalysis abnormal finding as defined in the Appendix to the protocol. Subjects with a Grade 1 biochemistry, hematology or urinalysis abnormality will be considered for inclusion on a case by case basis following discussion between the Investigator and the DMID Medical Monitor.
* Has any malignancy (excluding nonmelanotic skin cancer) or lymphoproliferative disorder diagnosed or treated actively during the past 5 years.
* A history or clinical evidence of hepatic disease, including abnormal laboratory values for AST, ALT or total bilirubin or abnormal laboratory values for potassium.
* A history or clinical evidence of hematological abnormalities; specifically abnormal laboratory values for hemoglobin, platelets, WBC or neutrophils.
* A history or clinical evidence of renal disease; specifically abnormal laboratory values for serum creatinine.
* A history or clinical evidence of ventricular arrhythmias, or any subject with an implantable defibrillator.
* A history or clinical evidence of significant respiratory disease (including asthma, hyper-reactive lung disease, COPD [on oral steroids or with chronic bronchitis], cystic fibrosis and/or recurrent lower respiratory tract infection, pneumonectomy or pulmonary insufficiency requiring home O2) and/or upper respiratory tract infection within the last 3 weeks or lower respiratory tract infection within the last 3 months.
* Any diagnosis of dementia (such as Alzheimer's disease) or current treatment for dementia (e.g. Aricept), or a mini mental state score of less than or equal to 25 at Screening.
* A Geriatric Depression Scale-Short Form (GDS-SF) score of greater than or equal to 6 (out of a total possible score of 15) at Screening, or a history or clinical evidence of endogenous depression, or a history or clinical evidence or treatment of exogenous depression within 1 year prior to enrollment in this study.
* A score of less than or equal to 16 out of 20 in the Clock Drawing Test (CDT) on Day 0.
* Has an acute or chronic medical condition that in the opinion of the Investigator would interfere with the evaluation of response.
* Is using parenteral or oral steroids, inhaled medications, anticoagulants, immune modulators (oral or topical) or other immunosuppressive or cytotoxic drugs within 2 weeks prior to enrolment in this study.
* Has received any other neuraminidase inhibitor within 2 weeks prior to enrollment in this study.
* A history or clinical evidence of dizziness with unknown cause.
* History of severe adverse reaction or hypersensitivity to lactose or neuraminidase inhibitors.
* Intake of any investigational drug product within 4 months prior to the intake of investigational product (Day 1).
* Receipt of blood or blood products or loss of 450 mL or more of blood during the last 3 months before screening.
* Has a clinically significant history of alcohol abuse or drug abuse.
* Body Mass Index (BMI) less than 18.5 kg/m2 or greater than 32.0 kg/m2.
* FEV1 less than or equal to 85%, FEV1.0% less than or equal to 70%, and/or FVC less than or equal to 80% of the predicted value, as calculated from standard age and height formula. If the first assessment is borderline then 2 further assessments may be made, both of which must have values above these criteria for the subject to be eligible.
* Subjects who smoke or have been non-smokers for less than 6 months prior to Screening.
* Subjects who were previously enrolled in this study.
* Poor veins or fear of venipuncture or sight of blood.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: treatment-emergent AEs, changes in vital signs including BP and PR, SpO2, oral body temperature, ECG, spirometry, PEFR, physical examinations, psychological assessments and laboratory parameters. | Duration of study

SECONDARY OUTCOMES:
Pharmacokinetic parameters for CS-8958 and R-125489. | Days 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Douglas ET Lee, MBChB MRCP DGM, Principal Investigator — Covance CRU
Locations (1):
- Covance Clinical Research Unit Ltd (Covance CRU), Leeds, United Kingdom